CLINICAL TRIAL: NCT06517771
Title: Online Aerobic Exercise During the COVID-19 Era: Exploring Physical Performance and Health-related Quality of Life Changes in Non-diagnosed COVID-19 Adults
Brief Title: Online Aerobic Exercise and Quality of Life in Non-diagnosed COVID-19 Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Gökhan Bayrak, Doctor Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 51099/8-45
Record Dates: First submitted 2024-07-22; First posted 2024-07-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online aerobic exercise group (Experimental): Participants in the online aerobic exercise group performed aerobic exercises three days a week for four weeks under the online supervision of a physiotherapist using the WhatsApp application.
  Interventions: Other: Online aerobic exercise
- Control group (No Intervention): The control group did not engage in any aerobic or strengthening exercise training during the four weeks and were instructed to avoid strenuous physical activities

INTERVENTIONS:
Other: Online aerobic exercise — Before starting the online aerobic exercises, for general warm-up, two minutes of walking, one minute of marching, and ten repetitions of bilateral reciprocal shoulder flexion-extension, shoulder horizontal abduction-adduction, and unilateral shoulder flexion and circling exercises were performed. For the upper extremity, full elbow extension with shoulder retraction in full shoulder flexion (Exercise V), elbows 90 degrees flexion with shoulder retraction in 90 degrees abduction (Exercise U), and full elbow flexion with shoulder extension of about 30 degrees (Exercise W) were performed. Standing hip abduction-extension, elevation on tiptoe, standing-sitting from a chair with hands on shoulders, squatting, tandem walking, and standing on one leg exercises were performed in the lower extremities. Gastrocnemius, hamstring, and shoulder posterior and inferior capsule stretching exercises were conducted as cooling exercises.
  Arms: Online aerobic exercise group

SUMMARY:
During the new coronavirus-19 (COVID-19) pandemic, assessing the effects of online aerobic exercise on physical performance and health-related quality of life (HRQoL) in adults has garnered significant interest. This study, which investigated the impact of four-week online aerobic exercise on physical performance and HRQoL in non-diagnosed COVID-19 adults, provides crucial insights. After the study was completed, the four-week online exercise program did not significantly enhance physical performance and HRQoL but increased physical activity. These findings are important for understanding the potential of online aerobic exercise. While it may not yield notable health-related benefits, it can boost physical activity in non-diagnosed COVID-19 adults.

DETAILED DESCRIPTION:
The rapid spread of the novel coronavirus disease-19 (COVID-19) pandemic has led clinicians to new and alternative methods and led the way for various practice strategies. Telehealth applications enable health professionals to transfer information, education, and training for health consumers via the Internet and telecommunication. Telehealth applications and remote assessment applications are technology and services that can be used during the COVID-19 pandemic process. In addition, practical applications can be made with the help of telephone and video in a guideline published concerning remote health applications.

The advantages of participation in exercise programs include improvements in physical performance, aerobic endurance, self-efficacy for exercise, self-assessed health, and pain relief. The COVID-19 pandemic has induced extensive disruptions to global health systems and accelerated the shift to remotely accessible counseling and home-based rehabilitation. Implementing remotely monitored exercise interventions has the advantages of greater access and accessibility and overcoming known barriers to face-to-face supervised exercise. In the COVID-19 pandemic, tele-exercise, including remote delivery of exercises via video conferencing technology, has emerged as a means for community-based programs to maintain follow-up exercise sessions while adhering to physical distancing restrictions. A previous investigation indicated that tele-yoga exercise sessions were feasible and acceptable in older adults. Social isolation, which required attention and practice during the COVID-19 pandemic, causes significant changes that negatively affect public health and physical activity levels. In the COVID-19 pandemic, remote exercise implementation methods mainly focused on patients with chronic diseases or the older population.

People who are not regularly active and have no contraindications are recommended to start and gradually increase their physical activity level. The World Health Organization guidelines for adults indicate that aerobic and muscle-strengthening physical activity exercises are based on solid evidence. Additionally, there needs to be randomized controlled studies in the literature regarding online physical exercise during COVID-19. Therefore, it is curious to evaluate the physical activity level and physical performance in adults during the COVID-19 pandemic and how exercise interventions will affect them. In this study, we aimed to examine the effect of online exercise training on physical performance and health-related quality of life (HRQoL) in non-diagnosed COVID-19 adults during the pandemic. As a hypothesis in our study, we hypothesized that four-week online exercise training would improve physical performance and HRQoL compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Not diagnosed with COVID-19,
* Being between 40-60 years of age,
* Having a medium level of physical activity according to the International Physical Activity Questionnaire-Short Form (IPAQ-SF),
* Not having any mental or physical problem preventing walking, running, or jumping,
* Residing in the Muş and Denizli city provinces,
* Being able to speak and understand the local language,
* Being able to understand verbal and written information given.

Exclusion Criteria:

* Having an injury/injury affecting the lower or upper extremities within the last six months,
* Participating in any exercise or strengthening training within the previous three months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | Baseline, Week 4
  The participants' physical activity levels were evaluated with the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The IPAQ-SF is a scale developed to determine the physical activity levels of participants aged 15-65 years and aims to obtain information about the time individuals spend in vigorous, moderate-to-vigorous activities and walking. The calculation of the IPAQ-SF total score includes the sum of the duration and frequency of walking, moderately vigorous, and vigorous activity in the last week. In physical activity level classification, individuals with a physical activity score of less than 600 Metabolic equivalents of task (MET) min/week are classified as low level, individuals with physical activity between 600-3000 MET min/week are classified as medium physical activity level, and individuals with physical activity more than 3000 MET min/week are classified as high physical activity level.
Physical Performance | Baseline, Week 4
  Short Physical Performance Battery (SPPB): The SPPB is calculated from three components: the ability to stand, time to complete a 3-m walk, and time to stand from a chair five times. Each part is scored out of 4, with the scores from the three tests calculated to give a total of 12 and a minimum of 0.
  Single-Leg Standing Test: For the single-leg participant stands in the dominant foot with the other knee at 90 degrees. If the participant reaches 30 seconds, the time is stopped.
  Four Square Step Test (FSST): For the FSST, the participant starts from a square with both feet, steps clockwise to the starting square, and returns to the starting square without stopping (start: right-back-left-front; return: back-right-front-left).
  Timed Up and Go (TUG) Test: For the TUG test, the participant has to get up from the chair, walk 3 meters, walk around the line on the floor, walk back to the chair, and sit down.
Health-Related Quality of Life | Baseline, Week 4
  The health-related quality of life (HRQoL) was evaluated with the Short Form-36 (SF36). SF-36 is a patient-reported questionnaire developed and used to determine HRQoL. It is a self-assessment scale with generic criteria. In this study, SF-36 physical function and general health subscales were utilized. The subscales assess health on a 0-100 scale, with 0 indicating poor health and 100 indicating good health

SECONDARY OUTCOMES:
Anxiety | Baseline, Week 4
  The Beck Anxiety Inventory (BAI) was utilized to evaluate the participants' anxiety levels. This self-report instrument comprises 21 items that assess subjective anxiety and physical symptoms, with each item scored on a Likert scale ranging from 0 to 3. The total score on the BAI can range from 0 to 63, with higher scores reflecting more severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Bayrak, PhD, Principal Investigator — Muş Alparslan University
Locations (1):
- Muş Alparslan University, Muş, Muş and Denizli Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not have a plan to make individual participant data available to other researchers

REFERENCES:
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] Canton-Martinez E, Renteria I, Machado-Parra JP, Reyes RA, Moncada-Jimenez J, Johnson DK, Gonzalez OM, Del Valle AS, Jimenez-Maldonado A. A virtually supervised exercise program improved fitness and mental wellness in healthy and comorbidity older adult individuals during the COVID-19 pandemic. Front Public Health. 2024 Apr 23;12:1328518. doi: 10.3389/fpubh.2024.1328518. eCollection 2024. PMID 38716241
- [Result] D'Oliveira A, De Souza LC, Langiano E, Falese L, Diotaiuti P, Vilarino GT, Andrade A. Home Physical Exercise Protocol for Older Adults, Applied Remotely During the COVID-19 Pandemic: Protocol for Randomized and Controlled Trial. Front Psychol. 2022 Feb 4;13:828495. doi: 10.3389/fpsyg.2022.828495. eCollection 2022. PMID 35185739
- [Derived] Bayrak G, Aslan UB. Four-week remotely supervised aerobic exercise during the COVID-19 era: Exploring physical performance and psychosocial health in adults without COVID-19 living in rural settings. Medicine (Baltimore). 2025 Aug 29;104(35):e44016. doi: 10.1097/MD.0000000000044016. PMID 40898552